CLINICAL TRIAL: NCT03212157
Title: Establishment of GlucoCEST MRI as a Biomarker in Cancer Translational Study
Brief Title: GlucoCEST MRI in Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 13/0450
Record Dates: First submitted 2017-06-27; First posted 2017-07-11 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Lymphoma; Glioma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoma; Glioma | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GT1 (Experimental): Optimsation of glucose infusion protocol outside the Magnetic Resonance Imaging (MRI) scanner in healthy volunteers. To establish an optimised bolus and safety of infusion protocol of intravenous glucose to maximise exchange sensitive MRI signal.
  Interventions: Other: Glucose infusion
- GT2 (Experimental): Optimsation of glucose infusion protocol inside the Magnetic Resonance Imaging (MRI) scanner in patient volunteers. To assess the reproducibility of these techniques and initial proof-of-concept study in cancer patients
  Interventions: Other: Glucose infusion; Diagnostic Test: Magnetic Resonance Imaging (MRI)
- GT3 (Experimental): Use of glucoCEST technique in staging of head and neck SCC, lymphoma and gliomas and correlating diagnostic potential with standard imaging such as FDG PET. To apply exchange-sensitive MRI in selected cancer types to assess its diagnostic potential. To study of non-glucose endogenous exchange sensitive MRI signals in (a) Prostate Cancer and (b) high grade Glioma patients.
  Interventions: Other: Glucose infusion; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: FDG PET

INTERVENTIONS:
Other: Glucose infusion — Infusion of 20% dextrose (drug) and using this as an imaging tracer in detecting and staging tumours.
Diagnostic Test: Magnetic Resonance Imaging (MRI) — MRI scanners (device) use strong magnetic fields, radio waves, and field gradients to generate images of the organs in the body. Specifically using the MRI scanner with the infusion of dextrose in detecting and staging tumours.
  Arms: GT2; GT3
Diagnostic Test: FDG PET — FDG is a sugar (glucose) labelled with a small amount of radioactivity which goes to parts of the body that use glucose for energy. PET/CT images are acquired on a single scanner. An FDG PET scan can be used to assess the presence, location and severity of cancers.
  Arms: GT3

SUMMARY:
The roles of imaging in cancer may be divided into that of diagnosis and tumour detection, staging and assessment of response to treatment. Standard radiological techniques include ultrasound, Computed Tomography (CT), Magnetic Resonance Imaging (MRI) and Positron Emission Tomography (PET). A combination of imaging techniques is often necessary to differentiate between cancerous and normal tissue. Traditional imaging techniques identify cancers by their gross appearance and structural/ cellular characteristics, whilst PET do so by tracking glucose metabolism. PET owes its specificity to the high rate of glucose metabolism seen in most cancers. However it is not used routinely due to a lack of availability and high costs. In addition, PET is often used in combination with CT, which imparts a significant diagnostic radiation dose. This can increase an individual's risk of cancer, especially with childhood or early adult exposure. In contrast, MRI is more readily available and does not involve radiation. However its ability to detect cancer by tracking glucose metabolism has not been widely explored. Our group has recently developed a novel MRI technique called Gluco-CEST that can image glucose delivery, uptake and metabolism in cancer, therefore potentially allowing a radiation-free, one-stop imaging service that can be adapted to current generation of MRI scanners. This study aims to optimise the GlucoCEST technique, after which it will be rigorously tested and compared to standard imaging parameters and clinical or pathological reference standards to evaluate its diagnostic and predictive power across a number of cancer populations.

DETAILED DESCRIPTION:
The technique involves administration of glucose solution either orally or intravenously. This is metabolised and concentrated into the intracellular compartment rapidly, which can be detected by GlucoCEST MRI. The abnormally high glucose uptake demonstrated by certain tumours is therefore potential biomarkers. At present this is already being investigated in head and neck cancer patients using oral glucose in a separate study. In this proposal we aim to utilise intravenous administration of glucose, which has been shown in pre-clinical studies to improve GlucoCEST signal, and thus likely to increase the detectability of cancer.

This study aims to develop and assess GlucoCEST and other exchange-sensitive MRI measurements (denoted 'exchange-sensitive MRI' hereafter) using intravenous glucose in tumours and metastases, and evaluate its use as an imaging biomarker of tumour and treatment response. This project will:

1. Establish an optimised bolus and infusion protocol of intravenous glucose to maximise exchange-sensitive MRI signal.
2. Assess the reproducibility of exchange-sensitive MRI and initial proof-of-concept study in cancer patients
3. Apply exchange-sensitive MRI in selected cancer types to assess its diagnostic and prognostic power.

The initial optimisation study involves investigating the optimal regime of intravenous glucose administration for obtaining the optimal exchange-sensitive MRI signal. The second stage will see exchange-sensitive MRI being applied to patients in different cancer groups to assess its ability for detecting cancer.

For the optimisation study, 20 healthy volunteers will be recruited. For the application study 80 patients (20 Hodgkin's lymphoma, 20 head and neck tumour, and 40 glioma) will be investigated. Most of these patients will be due for an MRI as part of their standard care pathway; in these cases exchange-sensitive MRI will be added to the standard imaging sequence. For those who are not otherwise due for MRI, both standard and exchange-sensitive MRI will be acquired.

It is expected that the data generated from this study will inform the design of larger trials and will provide the framework for an improved imaging pathway in certain cancer groups in the future.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers:

  1. No previous history of cancer
  2. No known renal impairment or an eGFR within a standard reference value if there is a history of renal disease.
  3. Aged 18 or over with capacity to consent.
* Patient groups:

  1. Confirmed diagnosis of selected cancer types (head and neck, lymphoma and glioma)
  2. No known renal impairment or an eGFR within a standard reference value if there is a history of renal disease
  3. Aged 18 or over with capacity to consent.

Exclusion Criteria:

* For both groups:

  1. Confirmed diagnosis of selected cancer types (head and neck, lymphoma and glioma)
  2. Pregnancy
  3. Contradiction to MRI magnetic field (pacemaker, metallic implant, severe claustrophobia, etc)
  4. Allergy to MR contrast agent (Gadolinium)
  5. Adult with Impaired capacity
  6. Deranged renal function with eGFR

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Developing new biochemical imaging tracer | 4 years
  Optimised exchange-sensitive MRI techniques using intravenous glucose. Evaluation of the added value of quantitative GlucoCEST imaging, derived using OM CEST analysis software, to standard multi-modality anatomical imaging
Assessing diagnostic value of glucoCEST | 4 years
  Exchange-sensitive MRI in selected cancer types to assess its potential diagnostic value. Pre-treatment and post-treatment quantitative GlucoCEST MRI will be evaluated for prediction of residual/recurrent disease against clinical outcome measures of DFS, TTP and OS.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker-Samuel S, Ramasawmy R, Torrealdea F, Rega M, Rajkumar V, Johnson SP, Richardson S, Goncalves M, Parkes HG, Arstad E, Thomas DL, Pedley RB, Lythgoe MF, Golay X. In vivo imaging of glucose uptake and metabolism in tumors. Nat Med. 2013 Aug;19(8):1067-72. doi: 10.1038/nm.3252. Epub 2013 Jul 7. PMID 23832090